CLINICAL TRIAL: NCT02068794
Title: Phase I/II Trial of Intraperitoneal Administration of Adipose Tissue Derived Mesenchymal Stem Cells Infected With a NIS-Expressing Derivative Manufactured From a Genetically Engineered Strain of Measles Virus in Patients With Recurrent Ovarian Cancer
Brief Title: MV-NIS Infected Mesenchymal Stem Cells in Treating Recurrent Ovarian, Primary Peritoneal or Fallopian Tube Cancer
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC1266; P50CA136393 (NIH); R01CA200507 (NIH); R01CA136547 (NIH); NCI-2014-00016 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1266 (Other: Mayo Clinic); 12-007859 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2014-02-19; First posted 2014-02-21 (Estimated); Results first posted 2025-07-16 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Fallopian Tube Clear Cell Adenocarcinoma; Fallopian Tube Endometrioid Adenocarcinoma; Fallopian Tube Mucinous Adenocarcinoma; Fallopian Tube Serous Adenocarcinoma; Fallopian Tube Transitional Cell Carcinoma; Fallopian Tube Undifferentiated Carcinoma; Malignant Ovarian Brenner Tumor; Ovarian Clear Cell Adenocarcinoma; Ovarian Endometrioid Adenocarcinoma; Ovarian Mucinous Adenocarcinoma; Ovarian Seromucinous Carcinoma; Ovarian Serous Adenocarcinoma; Ovarian Transitional Cell Carcinoma; Ovarian Undifferentiated Carcinoma; Primary Peritoneal Serous Adenocarcinoma; Recurrent Fallopian Tube Carcinoma; Recurrent Ovarian Carcinoma; Recurrent Primary Peritoneal Carcinoma
MeSH Terms: conditions — Brenner Tumor; Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — Mesenchymal Stem Cell Transplantation; Specimen Handling; X-Rays; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (MV-NIS infected mesenchymal stem cells) (Experimental): Patients receive oncolytic measles virus encoding thyroidal sodium iodide symporter IP over 30 minutes on day 1 of cycle 1 and MV-NIS infected MSC (if MSC are not available, MV-NIS may be given alone) IP over 30 minutes of subsequent cycles. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.
  Additionally, patients undergo ECHO or MUGA prior to registration and blood sample collection, chest X-ray, SPECT/CT, CT or MRI throughout the study.
  Interventions: Other: Laboratory Biomarker Analysis; Procedure: Mesenchymal Stem Cell Transplantation; Biological: Oncolytic Measles Virus Encoding Thyroidal Sodium Iodide Symporter; Procedure: Echocardiography; Procedure: Multigated Acquisition Scan; Procedure: Biospecimen Collection; Procedure: Chest Radiography; Procedure: Single Photon Tomography and Computed Tomography Scan; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Procedure: Mesenchymal Stem Cell Transplantation — Given IP
Biological: Oncolytic Measles Virus Encoding Thyroidal Sodium Iodide Symporter — Given IP
  Other Names: MV-NIS
Procedure: Echocardiography — Undergo ECHO
  Other Names: Echocardiograph (EC); echocardiograph; ECHO
Procedure: Multigated Acquisition Scan — Undergo MUGA
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide ventriculography; Radionuclide Ventriculography (RNVG); RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Blood Sample Collection; Specimen Collection
Procedure: Chest Radiography — Undergo chest X-ray
  Other Names: chest x-ray
Procedure: Single Photon Tomography and Computed Tomography Scan — Undergo SPECT/CT
  Other Names: SPECT/CT; SPECT/CT SCAN
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography (CAT); computerized axial tomography; Computerized axial tomography (procedure); Computerized Tomography; CT; CT SCAN; tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure)Q; Magnetic Resonance Imaging Scan; Medical Imaging; Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI Scan; MRIs; NMRI; nuclear magnetic resonance imaging; sMRI; Structural MRI

SUMMARY:
This phase I/II trial studies the side effects and best dose of oncolytic measles virus encoding thyroidal sodium iodide symporter (MV-NIS) infected mesenchymal stem cells and to see how well it works in treating patients with ovarian, primary peritoneal or fallopian tube cancer that has come back. Mesenchymal stem cells may be able to carry tumor-killing substances directly to ovarian, primary peritoneal and fallopian tube cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximally tolerated dose (MTD) of intraperitoneal administration of an Edmonston's strain measles virus genetically engineered to produce sodium iodine symporter (NIS) (measles virus [MV]-NIS) in patients with recurrent ovarian cancer, delivered by adipose tissue derived mesenchymal stem cells (MSC). (Phase I) II. To assess the 12 month overall survival of patients treated with this regimen. (Phase II)

SECONDARY OBJECTIVES:

I. To assess the tolerability of this regimen. (Phase II) II. To assess the 4 month progression free survival of patients treated with this regimen. (Phase II) III. To assess the response rate, progression-free survival, and overall survival of patients treated with this regimen. (Phase II)

TRANSLATIONAL OBJECTIVES:

I. To assess the time course of viral gene expression and virus elimination and biodistribution of virally infected cells at various time points after infection with MV-NIS versus MSC delivered MV-NIS using single-photon emission computed tomography (SPECT)/computed tomography (CT) imaging. (Phase II) II. To assess viremia, viral replication, and measles virus shedding/persistence following intraperitoneal administration. (Phase II) III. To assess humoral and cellular immune response to the injected virus. (Phase II) IV. To assess in a preliminary fashion the development of antitumor immune response. (Phase II)

OUTLINE: This is a phase I, dose-escalation study followed by phase II study.

Patients receive oncolytic measles virus encoding thyroidal sodium iodide symporter intraperitoneally (IP) over 30 minutes on day 1 of cycle 1 and MV-NIS infected mesenchymal stem cells (MSC) (if MSC are not available, MV-NIS may be given alone) IP over 30 minutes of subsequent cycles. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo echocardiography (ECHO) or multigated acquisition scan (MUGA) prior to registration and blood sample collection, chest X-ray, SPECT/CT, CT or magnetic resonance imaging (MRI) throughout the study.

After completion of study treatment, patients are followed up every 6 months for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Must have:

  * Recurrent or progressive ovarian cancer, primary peritoneal cancer or fallopian tube cancer after prior treatment with platinum and taxanes
  * Histologic confirmation of the original primary tumor
  * Prior bilateral oophorectomy
* The following histologic epithelial cell types are eligible: serous adenocarcinoma, endometrioid adenocarcinoma, mucinous adenocarcinoma, undifferentiated carcinoma, clear cell adenocarcinoma, mixed epithelial carcinoma, transitional cell carcinoma, malignant Brenner's tumor, or adenocarcinoma not otherwise specified (NOS)
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1, 2
* Absolute neutrophil count (ANC) >= 1500/uL (obtained =< 7 days prior to registration)
* Platelet (PLT) >= 100,000/uL (obtained =< 7 days prior to registration)
* Total bilirubin =< upper normal limit (obtained =< 7 days prior to registration)
* Aspartate aminotransferase (AST) =< 2 x upper limit of normal (ULN) (obtained =< 7 days prior to registration)
* Creatinine =< 1.5 x ULN (obtained =< 7 days prior to registration)
* Hemoglobin (Hgb) >= 9.0 g/dL (obtained =< 7 days prior to registration)
* Normal cardiac function as defined by a normal ejection fraction by MUGA (multi gated acquisition scan) or echocardiogram
* Provide informed written consent
* Willing to return to Mayo Clinic Rochester for follow-up
* Life expectancy >= 12 weeks
* Willing to provide all biologic specimens as required by the protocol
* Measurable disease by exam or CT scan, or for patients with cancer antigen (CA)-125 elevation or with microscopic residual but without measurable disease on imaging, willingness to undergo laparoscopy for evaluation of treatment effect if no radiographic progression after 6 treatment cycles
* CD4 count >= 200/uL or >= 15% of peripheral blood lymphocytes

Exclusion Criteria:

* Epithelial tumors of low malignant potential, stromal tumors, and germ cell tumors of the ovary
* Known standard therapy for the patient's disease that is potentially curative or definitely capable of extending life expectancy; subjects will be excluded if this is their first relapse and they have recurred > 6 months from completion of primary (adjuvant) chemotherapy
* Active infection =< 5 days prior to registration
* History of tuberculosis or history of tuberculosis skin test purified protein derivative (PPD) positivity
* History of other malignancy =< 5 years prior to registration except for non-melanoma skin cancer, carcinoma in situ of the cervix, and ductal carcinoma in situ (DCIS)
* Any of the following prior therapies:

  * Chemotherapy =< 3 weeks prior to registration
  * Immunotherapy =< 4 weeks prior to registration
  * Biologic therapy =< 4 weeks prior to registration
  * Extensive abdominal surgery if it includes enterotomy(ies) =< 3 weeks prior to registration; this criterion does not apply to placement of the peritoneal Port-A-Cath or lysis of adhesions at the time of registration
  * Any viral or gene therapy prior to registration
  * Radiation therapy to the abdomen or pelvis
* New York Heart Association classification III or IV, known symptomatic coronary artery disease, or symptoms of coronary artery disease on systems review, or known cardiac arrhythmias (atrial fibrillation or supraventricular tachycardia [SVT])
* Other cardiac or pulmonary disease that, at the investigators discretion, can impair treatment safety
* Requiring blood product support
* Central nervous system (CNS) metastases or seizure disorder
* Human immunodeficiency virus (HIV)-positive test result or history of other immunodeficiency
* History of organ transplantation
* History of chronic hepatitis B or C
* Other concurrent chemotherapy, immunotherapy, radiotherapy, or any ancillary therapy considered investigational (utilized for a non-Food and Drug Administration [FDA]-approved indication and in the context of a research investigation)
* Intra-abdominal disease > 8 cm in diameter at the time of registration, intrahepatic disease, or disease beyond the abdominal cavity; patients with intra-abdominal lymph node involvement are eligible based on biodistribution data indicating viral dissemination to lymph nodes following intraperitoneal administration
* Treatment with oral/systemic corticosteroids, with the exception of topical or inhaled steroids
* Exposure to household contacts =< 15 months old or household contact with known immunodeficiency
* Allergy to measles vaccine or history of severe reaction to prior measles vaccination
* Allergy to iodine; this does not include reactions to intravenous contrast materials
* Any other pathology or condition where the principle investigator may deem to negatively impact treatment safety

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2014-04-25 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2026-09-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Evanthia Galanis, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I Dose Level 0: Patients receive oncolytic measles virus encoding thyroidal sodium iodide symporter IP over 30 minutes on day 1 of cycle 1 and 10^7 MV-NIS infected MSC (if MSC are not available, MV-NIS may be given alone) IP over 30 minutes of subsequent cycles. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo ECHO or MUGA prior to registration and blood sample collection, chest X-ray, SPECT/CT, CT or MRI throughout the study.
- Phase I Dose Level 1; Phase II (Dose Level 1): Patients receive oncolytic measles virus encoding thyroidal sodium iodide symporter IP over 30 minutes on day 1 of cycle 1 and 10^8 MV-NIS infected MSC (if MSC are not available, MV-NIS may be given alone) IP over 30 minutes of subsequent cycles. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo ECHO or MUGA prior to registration and blood sample collection, chest X-ray, SPECT/CT, CT or MRI throughout the study.
Period: Overall Study
Arm/Group | Phase I Dose Level 0 | Phase I Dose Level 1 | Phase II (Dose Level 1)
Started | 4 | 7 | 23
Completed | 3 | 6 | 19
Not Completed | 1 | 1 | 4
Not completed — Withdrawal by Subject | 0 | 1 | 2
Not completed — Early Progression | 1 | 0 | 1
Not completed — Ineligible | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All eligible patients that completed at least one full cycle of treatment and monitoring.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I Dose Level 0 | Phase I Dose Level 1 | Phase II (Dose Level 1) | Total
Number analyzed (Participants) | 3 | 6 | 20 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.3 (12.74) | 62.3 (9.11) | 62.5 (8.94) | 62.1 (9.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 20 | 29
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 3 | 6 | 18 | 27
  Unknown or Not Reported | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 3 | 5 | 18 | 26
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Count of Participants That Experience a DLT
Description: Maximum tolerated dose will be defined as the dose level below the lowest dose that induces dose-limiting toxicity (DLT) in at least one-third of patients (at least 2 of a maximum of 6 new patients).
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I Dose Level 0 | Phase I Dose Level 1
Number analyzed (Participants) | 3 | 6
Participants | 0 | 0

2. Primary Outcome: Overall Survival at 12 Months
Description: The proportion of patients that were followed and alive at 12 months post registration.
Time Frame: 12 months
Population: Both Phase I and Phase II patients treated at dose level 1 are evaluable for this endpoint.
Measure: Number; unit: Proportion of patients
Groups:
- Phase I and II (Dose Level 1): Patients receive oncolytic measles virus encoding thyroidal sodium iodide symporter IP over 30 minutes on day 1 of cycle 1 and 10^8 MV-NIS infected MSC (if MSC are not available, MV-NIS may be given alone) IP over 30 minutes of subsequent cycles. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo ECHO or MUGA prior to registration and blood sample collection, chest X-ray, SPECT/CT, CT or MRI throughout the study.
Arm/Group | Phase I and II (Dose Level 1)
Number analyzed (Participants) | 26
Proportion of patients | 0.692

3. Secondary Outcome: Tumor Response (Phase II)
Description: Will be defined as complete response or partial response.
Time Frame: Up to 5 years
Reporting Status: Not Posted

4. Secondary Outcome: 4 Month Progression Free Survival Rate
Description: Defined as the proportion of patients alive and progression free at 4 months.
Time Frame: 4 months
Population: All evaluable patients treated at the maximum tolerated dose(Dose level 1) will be included in this analysis.
Measure: Number; unit: proportion of patients
Arm/Group | Phase I and II (Dose Level 1)
Number analyzed (Participants) | 26
proportion of patients | 0.769

5. Secondary Outcome: Overall Survival (Phase II)
Description: Defined as the length of time from study registration to date of death due to any cause. The distribution of survival time will be estimated using Kaplan-Meier survival curves and logrank tests.
Time Frame: Up to 5 years
Reporting Status: Not Posted

6. Secondary Outcome: Progression Free Survival (Phase II)
Description: Progression-free survival (PFS) is defined as the length of time from study registration to the first of either death due to any cause or progression. The distribution of PFS will be estimated using Kaplan-Meier survival curves and logrank tests. In addition, comparisons of overall PFS in patients treated with MV-NIS/MSC will be made to patients enrolled on the prior MV-CEA and MV-NIS trial in an exploratory manner.
Time Frame: Up to 5 years
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Time Course of Viral Gene Expression (Phase II)
Description: Descriptive statistics and simple scatterplots will form the basis of presentation of these data. Correlations between these laboratory values and other outcome measures will be carried out using Spearman's coefficients, chi squared tests, Wilcoxon rank-sum tests, Kaplan-Meier curves, and Cox proportional hazards models, where appropriate.
Time Frame: Up to 5 years
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Virus Elimination and Biodistribution of Virally Infected Cells by Single Photon Emission Computed Tomography Imaging (Phase II)
Description: as for outcome 7
Time Frame: Up to 5 years
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Incidence of Viremia (Phase II)
Description: as for outcome 7
Time Frame: Up to 5 years
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Incidence of Viral Replication (Phase II)
Description: as for outcome 7
Time Frame: Up to 5 years
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Measles Virus Shedding/Persistence Following Intraperitoneal Administration (Phase II)
Description: as for outcome 7
Time Frame: Up to 5 years
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Humoral Immune Response to the Injected Virus (Phase II)
Description: as for outcome 7
Time Frame: Up to 5 years
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Cellular Immune Response to the Injected Virus (Phase II)
Description: as for outcome 7
Time Frame: Up to 5 years
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Antitumor Immune Response (Phase II)
Description: as for outcome 7
Time Frame: Up to 5 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were followed for 8 months and mortality was followed for 5 years.
Arm/Group | Phase I Dose Level 0 | Phase I Dose Level 1 | Phase II (Dose Level 1)
All-Cause Mortality (participants affected / at risk) | 4/4 | 5/7 | 14/23
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/7 | 4/23
Other Adverse Events (participants affected / at risk) | 4/4 | 6/7 | 20/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I Dose Level 0 (N=4) | Phase I Dose Level 1 (N=7) | Phase II (Dose Level 1) (N=23)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3)
Infections and infestations - Oth spec (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I Dose Level 0 (N=4) | Phase I Dose Level 1 (N=7) | Phase II (Dose Level 1) (N=23)
Abdominal pain (Gastrointestinal disorders) | 2 (4) | 4 (8) | 16 (31)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 3 (5) | 9 (14)
Flatulence (Gastrointestinal disorders) | 0 (0) | 6 (21) | 7 (12)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (5) | 6 (7)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (3) | 5 (5)
Chills (General disorders) | 2 (4) | 2 (8) | 4 (6)
Fatigue (General disorders) | 0 (0) | 1 (3) | 3 (4)
Fever (General disorders) | 2 (4) | 1 (4) | 6 (7)
Activated partial throm time prolonged (Investigations) | 0 (0) | 0 (0) | 2 (3)
Alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 4 (7)
Neutrophil count decreased (Investigations) | 1 (1) | 1 (2) | 4 (4)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 6 (12)
White blood cell decreased (Investigations) | 0 (0) | 2 (3) | 6 (7)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 8 (11)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-03-22): https://cdn.clinicaltrials.gov/large-docs/94/NCT02068794/Prot_SAP_000.pdf
  • Informed Consent Form (2024-05-23): https://cdn.clinicaltrials.gov/large-docs/94/NCT02068794/ICF_001.pdf